CLINICAL TRIAL: NCT01812161
Title: Effect of Low-frequency Electroacupuncture (EA) on Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Heilongjiang University of Chinese Medicine (Other); Hubei College of Traditional Chinese Medicine (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dongmei Huang, Department of Integrated Traditional Chinese and Western Medicine Tongji hospital, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15002738313766868351
Record Dates: First submitted 2012-12-24; First posted 2013-03-18 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Electro-acupuncture; HCG stimulation test; Menstrual frequency; polycystic ovary syndrome; Randomized; controlled; trial
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture protocol 1 (Active Comparator): Acupuncture protocol 1：participants will receive treatment (acupuncture protocol 1, real acupuncture) twice a week; each treatment session can be separated by an interval of 2-4 days, with a maximum of 32 treatment sessions during 16 weeks. Each treatment session lasts for 30 minutes.
  Interventions: Other: acupuncture protocol 1
- Acupuncture protocol 2 (Sham Comparator): Acupuncture protocol 2：participants will receive treatment (acupuncture protocol 2, sham acupuncture) twice a week; each treatment session can be separated by an interval of 2-4 days, with a maximum of 32 treatment sessions during 16 weeks. Each treatment session lasts for 30 minutes. All participants will receive treatment twice a week; each treatment session can be separated by an interval of 2-4 days, with a maximum of 32 treatment sessions during 16 weeks. Each treatment session lasts for 30 minutes.
  Interventions: Other: Acupuncture protocol 2

INTERVENTIONS:
Other: acupuncture protocol 1 — Disposable, single-use, sterilized needles made of stainless steel, 0.25 x 30 mm and 0.30 x 40/50mm (Wuxi Jiajian Medical Instrument. 251226 Wuxi, China) will be inserted to a depth of 15-35 mm in some acupoints. After getting the needle sensation (de qi), some acupoints will receive electrical stimulation and the others will receive manual stimulation. All participants will receive treatment twice a week; each treatment session can be separated by an interval of 2-4 days, with a maximum of 32 treatment sessions during 16 weeks. Each treatment session lasts for 30 minutes.
  Other Names: real acupuncture
  Arms: Acupuncture protocol 1
Other: Acupuncture protocol 2 — Disposable, single-use, sterilized needles (0.20 x 20mm) made of stainless steel will be inserted to a depth of <5 mm at non-acupoints without evoking the needle sensation (Deqi). Electrodes will be attached to the needles and the stimulator will be turned on at an intensity of zero (no active current) in order to mimic EA in the acupuncture protocol 1 group. No manual stimulation of the needles will be performed.
  Other Names: sham acupuncture
  Arms: Acupuncture protocol 2

SUMMARY:
Low-frequency electroacupuncture (EA) can decrease serum 17-hydroxyprogesterone (17-OHP), androstenedione (A) and testosterone (T)of young women with polycystic ovary syndrome in the Human chorionic gonadotrophin (HCG) stimulation test ，also，we hypothesize that EA is more efficiency in improving ovulation rate and menstrual cycle than sham acupuncture.

DETAILED DESCRIPTION:
First, patients will be recruited according to the inclusion criteria and exclusion criteria.

Second, baseline measurements (including menstrual frequency,human chorionic gonadotropin (HCG) stimulation test,physical examination,trans-abdomen ultrasound of the uterus and ovaries, serum levels of sex hormone steroids) will be taken.

Third, each patient will receive 32 sessions of acupuncture in 16 weeks, twice a week.

Last, the above baseline measurements will be taken again as soon as the treatment is finished and menstrual frequency will be recorded during the 12 weeks of follow-up after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Unmarried women with age between 18 and 28 years and without bearing requirement within 4 months.
* 2) Confirmed diagnosis of PCOS according to the Rotterdam criteria: Oligomenorrhea(Menstrual cycle> 35 days, and less than 8 cycles per year), or amenorrhea (Menstrual cycle> 90 days) and one of the following two criteria; clinical or biochemical hyperandrogenism and/or polycystic ovarian morphology.

Exclusion Criteria:

* 1) Patients with hyperprolactinemia.
* 2) Patients with androgens secrete increased abnormal which caused by adrenal or ovarian tumors.
* 3) Patients with uncorrected thyroid disease[thyroid-stimulating hormone (TSH) <0.2 milli-International Unit /milliliter(mIU/mL) or >5.5 mIU/mL]except the patients with normal TSH in the past 1 year.
* 4)Suspected Cushing syndrome patients.
* 5)Patients who Received Estrogen, Progesterone or Oral contraceptives Oral contraceptives and hormone medications within the past 1 months. It takes at least one month to Eliminate these medicines, or it will influence the results
* 6) Patients who Received other medications that have influence on Reproductive function. or metabolism within the past 2 months( such as Anti obesity medications，Anti diabetic medications， traditional Chinese medicine and so on).
* 7)Patients who took acupuncture treatment within the past 3 months.
* 8)Patient who are unwilling to give written consent to the study.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
HCG stimulation test | 16 weeks
  Human chorionic gonadotrophin (HCG) stimulation test: Both at baseline and in one week after the treatment, the patients will receive an intramuscular injection of 5000 IU HCG, and 24 h and 48 h later, serum 17-hydroxyprogesterone (17-OHP), androstenedione (A) and testosterone (T) of the patients will be detected.

SECONDARY OUTCOMES:
Laboratory examination | 16 weeks
  Serum levels of sex hormone steroids including blood follicle-stimulating hormone (FSH), luteinizing hormone (LH), estrogen, progesterone, prolactin and total testosterone will be evaluated at baseline and 16 weeks. Oral glucose tolerance test (OGTT) and insulin releasing test will be performed at baseline and 16 weeks. Serum levels of leptin, adiponectin, resistin, adrenal cortical hormone and beta endorphin will be examined at baseline and 16 weeks later.
trans-abdomen ultrasound of the uterus and ovaries | 16 weeks
  The uterine dimensions, endometrial thickness and echo type, other uterine abnormalities, presence and size of leiomyoma, uterine artery blood flow parameters (pulsation index, resistance index, Shrinkage value / Diastolic value) will be obtained through trans-abdomen ultrasound at baseline and 16 weeks. The ovarian size in three dimensions, the size of the largest ovarian follicle/cyst and size of every follicle with a mean diameter greater than 10 mm, and total antral follicle (small follicles with mean diameter < 10 mm) count of each ovary; ovarian artery blood flow parameters will be observed through trans-abdomen ultrasound at baseline and 16 weeks later.
Physical examination | 16 weeks
  Physical examination including vital signs, height, weight, hip and waist measurements, BMI and assessment of hirsutism by Ferriman-Gallwey score and acne standard acne lesion counts will be performed at baseline and 16 weeks.
Number of Participants with Adverse Events | 16 weeks
  Adverse events happened during 16-week treatment period and 12-week follow-up will be recorded and classified. Unless otherwise formal requirements, each report about the detail and summary of adverse event to data safety supervision and the commission will be reported by double blind way.
menstrual frequency | 16 weeks
  The menstruation characteristics including menstrual cycle, duration and amount of the past 4 months and during the treatment period will be recorded. Menstrual frequency was calculated by dividing the number of menstrual bleeding by 4.
serum levels of the neurotransmitter | 16 weeks
  serum levels of AD, NE,5-HT and GABA between two groups both at baseline and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Huang, doctor, Principal Investigator — Department of Integrated Traditional Chinese and Western Medicine Tongji hospital of Huazhong University of Science and Technology
Locations (1):
- Department of Integrated Traditional Chinese and Western Medicine Tongji hospital of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
we use the Clinical Trial Management Public Platform to manage and share our date.
Supporting Information: CSR
Time Frame: September1th，2019，for 1 year
Access Criteria: only for research

REFERENCES:
- [Background] Jedel E, Labrie F, Oden A, Holm G, Nilsson L, Janson PO, Lind AK, Ohlsson C, Stener-Victorin E. Impact of electro-acupuncture and physical exercise on hyperandrogenism and oligo/amenorrhea in women with polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E37-45. doi: 10.1152/ajpendo.00495.2010. Epub 2010 Oct 13. PMID 20943753
- [Derived] Dong HX, Wang Q, Wang Z, Wu XK, Cheng L, Zhou ZM, Yang L, Yi P, Huang DM. Impact of Low Frequency Electro-acupuncture on Glucose and Lipid Metabolism in Unmarried PCOS Women: A Randomized Controlled Trial. Chin J Integr Med. 2021 Oct;27(10):737-743. doi: 10.1007/s11655-021-3482-z. Epub 2021 Jul 28. PMID 34319506
- [Derived] Wang Z, Dong H, Wang Q, Zhang L, Wu X, Zhou Z, Yang L, Huang D. Effects of electroacupuncture on anxiety and depression in unmarried patients with polycystic ovarian syndrome: secondary analysis of a pilot randomised controlled trial. Acupunct Med. 2019 Feb;37(1):40-46. doi: 10.1136/acupmed-2017-011615. Epub 2019 Mar 7. PMID 30843421